CLINICAL TRIAL: NCT03189602
Title: Pulmonary Artery Involvement in Takayasu's Arteritis: a Retrospective Study in China
Brief Title: Pulmonary Artery Involvement in Takayasu's Arteritis
Status: Completed | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PUMCH-Pulmonary arteritis
Record Dates: First submitted 2017-06-15; First posted 2017-06-16 (Actual); Last update posted 2017-06-16 (Actual); Status verified 2017-06

CONDITIONS: Takayasu Arteritis; Pulmonary Artery Hypertension
Keywords: Takayasu Arteritis; Pulmonary artery hypertension
MeSH Terms: conditions — Takayasu Arteritis; Familial Primary Pulmonary Hypertension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to analyze the clinical manifestations, imaging features, and prognosis-related factors of pulmonary artery (PA) involvement in Takayasu's arteritis (TA), and to explore the early clinical features of PA involvement in TA patients.

DETAILED DESCRIPTION:
Takayasu's arteritis patients with pulmonary artery involvement were enrolled into this study. The demographic information of the patients (age, sex, course of disease), symptoms at their admissions (cough, hemoptysis, dyspnea, palpitations, fever), laboratory examinations (blood lab routines, erythrocyte sedimentation rate, C-reactive protein), and imaging examinations (vascular ultrasonography, computed tomographic angiography, echocardiography, chest CT, CTPA, pulmonary perfusion imaging, pulmonary angiography, PET/CT) were collected by reviewing the cases. The prognostic information was collected by telephone follow-up. The follow-up end point was December 2015.

ELIGIBILITY:
Inclusion Criteria:

* 1.Meet the diagnostic criteria of TA as defined by the American College of Rheumatology (ACR).
* 2.PA involvement: meet at least one of three items: (1) at least one of computed tomographic pulmonary angiography (CTPA), pulmonary perfusion imaging, or pulmonary arteriography suggests thickening of vessel wall, stenosis, aneurysm, or occlusion; (2) 18F-fluorodeoxyglucose positron emission tomography/computed tomography (PET/CT) suggests high intake of local radioactive material in pulmonary artery wall; (3) pulmonary artery systolic blood pressure is higher than 50 mmHg assessed by transthoracic echocardiography (defined as PAH), without left ventricular disease.

Exclusion Criteria:

-

Ages: 14 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Takayasu's arteritis patients with pulmonary artery involvement
Sampling Method: Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
Pulmonary Artery Systolic Blood Pressure | 1day
  Pulmonary artery systolic blood pressure(PASP) assessed by transthoracic echocardiography when admission. PASP>50mmHg is defined as pulmonary hypertension.

CONTACTS AND LOCATIONS:
Overall Officials: Juhong Shi, M.D, Study Chair — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Yang J, Peng M, Shi J, Zheng W, Yu X. Pulmonary artery involvement in Takayasu's arteritis: diagnosis before pulmonary hypertension. BMC Pulm Med. 2019 Nov 27;19(1):225. doi: 10.1186/s12890-019-0983-7. PMID 31775708